CLINICAL TRIAL: NCT01228110
Title: Corticosteroids and ICU Course of Community Acquired Pneumonia in Egyptian Settings
Brief Title: Corticosteroids in Community Acquired Pneumonea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Emad El-Din Omar, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06111972
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2009-07

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corticosteroid group (Active Comparator): This group was entitled to receive hydrocortisone 200 mg loading bolus followed by an intravenous infusion (300 mg in 500 ml 0.9% saline) at a rate of 12.5 mg/hour for 7 days
  Interventions: Drug: Hydrocortison
- Placebo group (Placebo Comparator): This group was meant to receive placebo (sterile normal saline in a volume equal to the study drug).
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Hydrocortison
  Arms: Corticosteroid group
Drug: Saline Solution
  Arms: Placebo group

SUMMARY:
Low dose hydrocortisone IV in patients with CAP fastens recovery of pneumonia and prevents the development of sepsis related complications with a significant reduction in duration of mechanical ventilation

DETAILED DESCRIPTION:
Inclusion Criteria Minor criteria includes

* respiratory rate > 30 bpm at admission;
* ratio of PaO2 to fraction of inspired oxygen (PaO2:FIO2 ) < 250;
* chest radiograph showing bilateral involvement or multilobar involvement;
* systolic blood pressure < 90 mm Hg; or
* diastolic blood pressure < 60 mm Hg. Major criteria includes
* Requirement of MV;
* Increase in the size of opacities on chest radiograph of 50% or more at 48 hours;
* Requirement of vasopressors for more than 4 hours; or
* Serum creatinine 2 mg/dl or more.

Exclusion criteria:

* Children;
* Nosocomial pneumonia;
* Hospitalisation within the previous 14 days;
* Severe immunosuppression (chronic use of systemic steroids);
* Non-steroid immunosuppressive treatment or HIV);
* Chronic chest disease; , tuberculosis, aspiration or obstructive pneumonia;
* Congestive heart failure (cerebrovascular stroke);
* Chronic renal or hepatic disease;
* Acute burn injury;
* Malignancy;
* Pregnancy; and
* Major gastrointestinal bleed within 3 months of the current hospitalization

Study Outcome The end-points of the study were improvement in PaO2:FIO2 (PaO2:FIO2 > 300 or ≥100 increase from study entry) and sepsis related organ failure assessment, (SOFA) score by day 8 and the development of delayed septic shock.

The adopted SOFA score (up to 6 points) was proposed by Vincent et al., [21]. The number of MV-free days was defined as the number of days after ventilation was discontinued up to study day 8. Shock was defined as requirement of vasopressors. ARDS was defined by consensus criteria.

All the patients were subjected to

1. Routine laboratory screen, including CBC, RBS, serum urea and creatinine, liver enzymes, serum billirubin and coagulation profiles;
2. Chest X ray on at least on admission and at day 8;
3. ABG at least once daily to detect PaO2:FIO2;
4. CRP daily from day 1 to 8 and
5. Evaluation of SOFA score daily

ELIGIBILITY:
Inclusion Criteria:

Minor criteria included

* respiratory rate > 30 bpm at admission;
* ratio of PaO2 to fraction of inspired oxygen (PaO2:FIO2 ) < 250;
* chest radiograph showing bilateral involvement or multilobar involvement;
* systolic blood pressure < 90 mm Hg; or
* diastolic blood pressure < 60 mm Hg. Major criteria included
* Requirement of MV;
* Increase in the size of opacities on chest radiograph of 50% or more at 48 hours;
* Requirement of vasopressors for more than 4 hours; or
* Serum creatinine 2 mg/dl or more. 10

Exclusion Criteria:

* Children;
* Nosocomial pneumonia;
* Hospitalisation within the previous 14 days;
* Severe immunosuppression (chronic use of systemic steroids);
* Non-steroid immunosuppressive treatment or HIV);
* Chronic chest disease; , tuberculosis, aspiration or obstructive pneumonia;
* Congestive heart failure (cerebrovascular stroke);
* Chronic renal or hepatic disease;
* Acute burn injury;
* Malignancy;
* Pregnancy; and
* Major gastrointestinal bleed within 3 months of the current hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)

PRIMARY OUTCOMES:
PaO2:FIO2
  improvement in PaO2:FIO2 (PaO2:FIO2 > 300 or ≥100 increase from study entry) and sepsis related organ failure assessment, (SOFA) score by day 8 and the development of delayed septic shock.